CLINICAL TRIAL: NCT02794844
Title: Implementation of Pharmacogenomic Testing in Nemours Children's Health System
Brief Title: Implementation of PPI Medication PGX Testing
Acronym: PGX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, James Franciosi, Principle Research Scientist, Nemours Children's Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 744230
Record Dates: First submitted 2016-04-27; First posted 2016-06-09 (Estimated); Results first posted 2018-05-09 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-10

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Omeprazole; Esomeprazole; Lansoprazole; Proton Pump Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Genotype Guided PPI Dosing (Experimental): Genotype Guided PPI Dosing: PI type and dosing will be recommended in real time based on patients' CYP2C19 genotype / metabolizer phenotype.
  No other ARM will be studied.
  Interventions: Drug: Genotype Guided PPI Dosing

INTERVENTIONS:
Drug: Genotype Guided PPI Dosing — Dosing of PPIs such as Prevacid and Nexium will be recommended based on CYP2C19 genotype information.
  Other Names: Prilosec; Nexium; Prevacid; Proton Pump Inhibitor

SUMMARY:
Using genetic information about the individual to pick the right drug for the right disease at the right dose defines personalized medicine. This pilot study seeks to institute pharmacogenomic testing, that is identifying genetic variation that influences patient response to drugs, into the Nemours Children's Health system. We propose to initiate the study by identifying genetic differences in cyp2c19, a gene that is responsible for a certain enzyme in the liver that metabolizes many drugs including a class of drugs called proton pump inhibitors (ppi; Prevacid, Nexium). PPIs are used to treat heartburn and other symptoms of gastroesophageal reflux disease (gerd) and are extensively used in pediatrics. Chronic use of PPIs can cause serious side effects including cold, pneumonia and stomach infections, which gets worse at higher doses. Children who poorly metabolize drugs because of genetic variation in cyp2c19 should get lower doses of PPIs than children who metabolize PPIs normally. Our pilot study will genotype children with gerd or other stomach acid mediated conditions for which a PPI is prescribed using a sample of spit to determine which dose of PPI they get based on the form of the cyp2c19 gene they have. We will study 120 children 2-17 yo diagnosed with gastroesophageal reflux disease (gerd) or other stomach acid mediated conditions for which a ppi is prescribed . Genetic results are available in < 60 minutes, and their doses are determined by their doctor based on genetic results. This study will allow us to gain valuable experience that will be used to expand our genetic program to other genes and drugs.

DETAILED DESCRIPTION:
The long-term objective of this research is to implement pharmacogenomic (PGX) testing of approved gene-drug pairs to maximize the efficacy and minimize adverse events for drugs that are used to treat childhood disease. Personalized medicine, that is, the use of the patient's own genetic information to predict the right dose of the right drug, has been a goal of medicine's since the publication of the human genome and HAPMAP projects. However, the adoption of PGX testing has been slow owing to several barriers and challenges. Recently President Obama announced the precision medicine initiative, which includes PGX testing, and has earmarked $ 1 b to implement it. The precision medicine initiative is expected to move personalized medicine forward so that most patients including pediatric patients will benefit. The Nemours Children's Health System is uniquely positioned to lead the effort to personalize medicine among pediatric patients. The goal of the proposed 1-year pilot project is to implement PGX testing in the Nemours children's health system. The experience, knowledge and skills gained in this pilot project will position Nemours to help lead precision medicine initiatives including PGX testing among pediatric populations. To implement PGX testing in Nemours we propose to begin testing the cyp2c19 - proton pump inhibitor gene-drug pair in the division of gastroenterology, Nemours children's hospital. A total of 120 children 2-17 yo who have been diagnosed with gastroesophageal reflux disease (GERD) or other stomach acid mediated conditions for which a PPI is prescribed will be recruited into the study by pediatric gastroenterologists (aim 1a). Drs. Franciosi and Lima will educate staff in the division of PGX testing and of the study. GI pediatricians are not required to participate in PGX testing. After obtaining consent, the study coordinator will obtain and bar code samples of saliva from the patient. Samples will be genotyped by Spartan Rx, a point-of-care genotyping platform, which are housed (2 of them) in the division of pathology. Loss-of-function alleles (*2, *3) and the gain-of-function allele (*17) are identified in < 60 minutes. The result of genotyping will be checked by dr. Badizadegan and entered into the patient's EMR. Clinical Decision Support (CDS) tools will advise Drs. Badizadegan and Franciosi of the patient's metabolic phenotype based on cyp2c19 genotype. Dr. Franciosi (or other GI pediatricians) will decide the dose of PPI to use based CDS tools carrying algorithms for conventional dosing and for genotype-guided dosing of PPIs. The electronic prescription for the PPI with genotype-guided dosing will be called in. PPI efficacy and safety for each study participant will be monitored weekly (aim 1B) by collecting and recording scores on validated GERD and adverse reaction questionnaires. Efficacy and safety scores will be communicated by each participant (or caregiver) using mobile devices (iPhone; computer) and recorded using redcap. Dr. Blake will supervise this phase of the study. Outcome metrics for aim 1A include: % of patients agreeing to volunteer for the study; % of patients reporting efficacy and toxicity data; % of providers agreeing to participate in study; and % of participants agreeing to future use of DNA. Outcome metrics for aim B will be judgments by Dr. Franciosi and his staff regarding success based on scores from GERD and adverse event questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with Gastroesophageal Reflux Disease (GERD) or a stomach acid mediated condition for which a PPI is prescribed.
* Currently taking or will be prescribed Proton Pump Inhibitor (PPI) medication
* Parents/legal guardians and or child must also have access to the internet and a valid email address to complete weekly required forms.

Exclusion Criteria:

* Children who have had peptic ulcer surgery;
* with a history of PKU
* with a history of previous adverse effects from PPI treatment or a sensitivity to aspartame (NutraSweet, Equal);
* who are non-adherent including inability or unwillingness of the legal guardian to provide consent of unwillingness of the child to provide assent;
* who are unable to take study medications;
* who are unable to communicate via telephone or other device;
* who do not have access to a computer with internet access

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2016-07-21 (Actual); Primary Completion 2017-01-23 (Actual); Study Completion 2018-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James P Franciosi, MD, Principal Investigator — Nemours Children's Hospital
Locations (1):
- Nemours Children's Hospital, Orlando, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 06/16/2015 to 02/20/2017, patients (or in the case of children, the pediatric patient and their parent/legal guardian) were approached for participation after a clinical assessment was performed by a GI provider during an outpatient GI appointment. Study procedures were performed after obtaining proper consent and/or child assent.
Groups:
- Genotype Guided PPI Dosing: Genotype Guided PPI Dosing: PPI type and dosing will be recommended in real time based on patients' CYP2C19 genotype / metabolizer phenotype.
  No other ARM will be studied.
Period: Overall Study
Arm/Group | Genotype Guided PPI Dosing
Started | 28
Completed | 23
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Genotype Guided PPI Dosing
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 16
  More than one race | 0
  Unknown or Not Reported | 5
Metabolizer Phenotype Frequency [Count of Participants; unit: Participants] — Depending on the CYP2C19 genotype individuals are classified into different phenotypes: poor metabolizer (PM), intermediate metabolizers (IM), normal metabolizers (NM), rapid metabolizer (RM) and ultra-rapid metabolizers (UM).
  Allele Genotype/Activity Phenotype
  * 1/*1 -2 active alleles NM
  * 1/n -1 active, 1 LOF allele IM
  * 2/*2 or *n*n -2 LOF alleles PM
  * 1/*17 -1 active, 1 GOF allele RM
  * 17/*17 -2 GOF alleles UM Population: Results were inconclusive for 5 participants
  Participants
    number analyzed (Participants) | 23
    Slow Metabolizers (IM and PM) | 5
    Normal Metabolizers (NM) | 11
    Fast Metabolizers (EM and UM) | 7

OUTCOME MEASURES:

1. Primary Outcome: Count of Patients Agreeing to Volunteer for the Study
Description: Outcomes for evaluating the success of PGX implementation
Time Frame: Through 12 months study
Measure: Count of Participants; unit: Participants
Groups:
- Genotype Guided PPI Dosing: Genotype Guided PPI Dosing: PI type and dosing will be recommended in real time based on patients' CYP2C19 genotype / metabolizer phenotype.
  No other ARM will be studied.
  Genotype Guided PPI Dosing: Dosing of PPIs such as Prevacid and Nexium will be recommended based on CYP2C19 genotype information.
Arm/Group | Genotype Guided PPI Dosing
Number analyzed (Participants) | 28
Participants | 28

2. Primary Outcome: Count of Patients Reporting Efficacy and Toxicity Data
Description: Outcomes for evaluating the success of PGX implementation
Time Frame: Throughout 12 month study
Measure: Count of Participants; unit: Participants
Arm/Group | Genotype Guided PPI Dosing
Number analyzed (Participants) | 28
Participants | 28

3. Primary Outcome: Count of Providers Agreeing to Participate in Study
Description: Outcomes for evaluating the success of PGX implementation
Time Frame: Throughout 12 month study
Population: 6 providers participated in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Genotype Guided PPI Dosing
Number analyzed (Participants) | 6
Participants | 6

4. Primary Outcome: Count of Participants Agreeing to Future Use of DNA
Description: Outcomes for evaluating the success of PGX implementation
Time Frame: Throughout 12 month study
Measure: Count of Participants; unit: Participants
Arm/Group | Genotype Guided PPI Dosing
Number analyzed (Participants) | 28
Participants | 28

5. Primary Outcome: Adverse Effects After Genotype-guided PPI Therapy
Description: Count of participants reporting adverse effects after genotype-guided PPI therapy.
Time Frame: Throughout 12 month study
Measure: Count of Participants; unit: Participants
Arm/Group | Genotype Guided PPI Dosing
Number analyzed (Participants) | 28
Participants | 11

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Genotype Guided PPI Dosing
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 11/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Genotype Guided PPI Dosing (N=28)
Sore Throat (Gastrointestinal disorders) | 6 (6)
Cold (Infections and infestations) | 7 (7)
Ear Infection (Infections and infestations) | 1 (1)
Sinus Infection (Infections and infestations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-10): https://cdn.clinicaltrials.gov/large-docs/44/NCT02794844/Prot_SAP_001.pdf